CLINICAL TRIAL: NCT06025565
Title: Measuring Pain Experience in Individuals With Lateral Elbow Tendinopathy
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: iRISID-2023-1767
Record Dates: First submitted 2023-08-18; First posted 2023-09-06 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Elbow Tendinopathy; Tendinopathy; Tennis Elbow
Keywords: Pain
MeSH Terms: conditions — Elbow Tendinopathy; Tendinopathy; Tennis Elbow; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LET: Patients with tennis elbow.
  Interventions: Diagnostic Test: Pain Experience Measures

INTERVENTIONS:
Diagnostic Test: Pain Experience Measures — Patient reported outcomes measures, quantitative sensory testing, and physical examination measures.

SUMMARY:
The study will address the gaps in the pain experience measurement in those with lateral elbow tendinopathy (LET) by building on the current body of literature, as well as applying modern pain science measures. The comprehensive measurement of various biomedical, psychological, and psychosocial constructs will provide pain profiles that will allow for the subclassification of LET to better inform loading prescriptions based on the systemic effects from LET.

DETAILED DESCRIPTION:
Methods: Subjects complete the eight patient reported questionnaires as well as go through 4 clinical examination procedures. Through this cross-sectional design and single session of testing, the investigator seeks to identify associations amongst constructs and variables in order to sub classify patients with LET based on their pain experience.

Study aim 1: The goal of this study is to determine the associations among the various measurements of the pain experience, psychological, psychosocial, and biomedical domains in those with LET.

Research Questions

1. How is the pain experience in individuals with LET associated with chance locus of control (LOC)?
2. What is the impact of fear avoidance on the pain experience in those with LET?
3. How does central sensitization alter the pain experience in those with LET?
4. Which pain experience measures are associated with functional ability in LET?

Hypotheses

1. Individuals with chance locus of control (LOC) will exhibit an increase in pain experience measures.
2. Individuals with fear avoidance will have an increase in pain experience measures.
3. Individuals with central sensitization (central sensitization inventory (CSI) > 40) will have an increase in pain experience measures.
4. Pain-free grip strength will have the largest positive correlation with patient-specific functional scale.

Background and Significance

Lateral elbow tendinopathy (LET) is a condition characterized by pain limiting upper extremity function that is not always easily managed, underscoring limits in the understanding and application of pain science. The problems with conservative management of LET appear to be rooted in the understudied and underutilized measurement of pain experience. This lack of research in the application of pain science in those with LET presents an opportunity when determining the appropriate loading of an injured tendon based on different subclassifications.

The complexity of tendinopathy pathogenesis and individual factors influencing the pain experience in those with LET requires a comprehensive series of measures to investigate what is unknown in this area. The use of novel or minimally investigated pain classification and psychological measures will provide insight into their influence on the pain experience to assist with subclassification. Quantitative sensory test (QST) gold standard tests (PPT and PFGS), as well as emerging tests (TPD and laterality), will provide clinical tests that may impact the pain experience and further support the current systematic theoretical mechanisms of tendinopathy. Using a cross-sectional study design will allow for higher recruitment numbers and improve the feasibility of the study. The investigator will investigate the known challenges in the pain measurement of LET and explore how they contribute to the lack of optimal loading in those with LET with respect to the biomedical, psychological, and psychosocial domains.

Subjects will be recruited from clinics in the Philadelphia, PA region. Convenience sampling will be employed through clinical staff to identify eligible subjects using the inclusion and exclusion criteria below. Recruitment will be through flyers and the Office of Recruitment Enhancement services at Thomas Jefferson University utilizing electronic medical record system notifications and emails. Subjects will be screened for eligibility and, if willing to participate, be provided informed consent by the investigator before participation.

Subjects will provide demographic information, and all patient-reported outcome measures (Patient-Specific Functional Scale (PSFS), Numeric Pain Rating Scale (NPRS), Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2), Central Sensitization Inventory (CSI), Multidimensional Health Locus of Control-C (MHLOC), Pain Catastrophizing Scale (PCS), Fear Avoidance Belief Questionnaire (FABQ), and Hospital Anxiety and Depression Scale (HADS). Subjects will then be tested on the physical measures (Two-Point Discrimination (TPD), Pressure Pain Threshold (PPT), Pain-Free Grip Strength (PFGS), and Laterality).

ELIGIBILITY:
Inclusion Criteria:

* English speaking and reading
* Aged 18-75
* Diagnosis of lateral elbow tendinopathy provoked by 2 clinical tests: painful resisted 2nd or 3rd finger extension, painful wrist extension, painful stretching of forearm extensor muscles, or painful gripping.

Exclusion Criteria:

* Receiving any medical intervention for LET from a physician within 90 days. Medical intervention operationally defined as any intervention requiring a medical state license to administer (injection or surgery) or prescribe (medication applied to or ingested that is not available without a physician script) with the exception of patient education.
* Positive mechanical sensitivity of the median nerve (Upper Limb Tension Test a (ULTTa)).
* Positive pain provocation of passive elbow flexion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient orthopedic clinics and those located throughout the Philadelphia region.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-08-18 (Actual); Primary Completion 2025-06-14 (Actual); Study Completion 2025-06-14 (Actual)

PRIMARY OUTCOMES:
Short Form-McGill Pain Questionnaire-2 | Baseline
  1. The subject will be asked to rate their pain on a 0-10 scale for 22 different pain descriptors.
  2. Continuous (1, 5, 6, 8, 9, 10), Intermittent (2, 3, 4, 11, 16, 18), Neuropathic (7, 17, 19, 20, 21, 22), and Affective (12, 13, 14, 15) subscales will be calculated by taking the mean of these items scores in addition to total score.
  3. The subject will also mark their pain on a numeric pain rating score.
  4. Scale is 0-10.
  5. Higher score is worse.
Patient Specific Functional Scale | Baseline
  1. The subject will identify 3 activities that are most limited and meaningful to them.
  2. The subject will rate these activities on an 11-point scale ranging from 0 "unable to perform" to 10 "Able to perform the activity at the same level as before the injury or problem."
  3. Scale is 0-30.
  4. Higher score is better.
Central Sensitization Inventory | Baseline
  1. The subject will be asked to assess for the presence of a central sensitization state on 25 questions scored in ordinal fashion 0 (never) - 4 (always).
  2. Data from this instrument will be obtained by recording the total score on a scale of 0-100.
  3. Higher score is worse.
Multidimensional health locus of control scale form C | Baseline
  1. The subject rates their opinion or sense that his/her outcomes are determined by luck, fate, or a random occurrence that controls experiences.
  2. The 6-point Likert scale is rated from strongly agree to strongly disagree, with 18 questions with 3 subscales including different types of loci of control (LOC; internal, chance, and doctors).
  3. Chance LOC scores range from 6-36 in an ordinal measurement.
  4. Data from this instrument will be obtained by recording the total score on a scale of 6-36.
  5. Higher score is worse.
Pain Catastrophizing Scale | Baseline
  1. The subject will be asked to assess for the presence of a pain catastrophizing on 13 questions scored in ordinal fashion 0 (not at all) - 4 (all the time).
  2. Data from this instrument will be obtained by recording the total score on a scale of 0-52.
  3. Higher score is worse.
Fear Avoidance Belief Questionnaire | Baseline
  1. The subject will be asked to assess for the presence of fear avoidance behavior.
  2. Items are scored on a 6-point Likert scale with questions 2-5 a subscale for work and 6, 7, 9, 10, 11, 12, and 15 for physical activity.
  3. Scale is 0-66.
  4. Higher score is worse.
Hospital Anxiety and Depression Scale | Baseline
  1. The subject will be asked to assess for the presence of anxiety or depression on 14 questions scored in 4-point Likert scale.
  2. Data from this instrument will be obtained by recording the total score and subscores for anxiety and depression.
  3. Scale is 0-56
  4. Higher score is worse.

SECONDARY OUTCOMES:
Pressure Pain Threshold | Baseline
  1. The subject will be seated with their affected arm positioned in a comfortable, relaxed position on the armrest of a chair.
  2. The Commander Echo Algometer will be used to assess the amount of pressure that can be applied at the lateral epicondyle before the onset of pain. The applicator (1 cm) will be positioned over the insertion of the forearm musculature at the lateral epicondyle.
  3. The subject will be instructed to verbally indicate when the pain begins by saying "stop."
  4. The tester will gradually apply an increasing amount of force at 1kg/second until the subject says "stop." This measure will be taken 3x in an alternating manner, in both arms, starting with the left with a 15 second rest between tests.
Two Point Discrimination | Baseline
  1. Affected elbow will be tested with two point discrimination.
  2. Subject will be seated in a neutral position with the elbow resting on the arm of a chair.
  3. Subjects will be asked to close their eyes to avoid additional stimulus and input.
  4. Calipers will be applied with pressure sufficient to blanch skin along the extensor mass of the elbow.
  5. The subject will report after each application "one", if one point is felt or "two", if two points are felt.
  6. If unsure, the subject is to report one point.
  7. Assessment will begin at 20 mm. The distance between the two points will gradually increase by 1 mm until the subject discerns two points.
  8. The distance that the subject first reports two points will be recorded.
  9. Measures will be take in both elbows.
Laterality | Baseline
  1. Subject will be seated and given a handheld device to hold.
  2. The subject will be instructed to review the images on the screen and as quickly and as accurately as they can, select whether the upper extremity on the screen is either left or right.
  3. The subject will complete the test after 25 images and the speed (seconds) and accuracy (%) of the test will be reported.
Pain-Free Grip Strength | Baseline
  1. In a seated position with the affected elbow flexed to 90º and wrist in a neutral position, the subject squeezes the Commander Echo Wireless Grip Strength tester as hard as they can until their elbow pain is reproduced.
  2. This procedure will be conducted at each rung position until the grip reproduces the subject's pain. Once the point of a painful grip is reached, the subject can rest for 30 seconds before testing.
  3. Subjects will be taken through painful grip testing 3x in each hand in an alternating manner with 15 second breaks between attempts starting in the left hand.
  4. Each painful grip measure of kg will be recorded

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Philadelphia Hand to Shoulder Clinic, Cape May, New Jersey
  - Philadelphia Hand to Shoulder Center, Cherry Hill, New Jersey
  - Philadelphia Hand to Shoulder Center, Collegeville, Pennsylvania
  - Jefferson Rehabilitation, Fairless Hills, Pennsylvania
  - Philadelphia Hand to Shoulder Center, Glen Mills, Pennsylvania
  - Philadelphia Hand to Shoulder Center, King of Prussia, Pennsylvania
  - Philadelphia Hand to Shoulder Center, Langhorne, Pennsylvania
  - Philadelphia Hand to Shoulder Center, Lansdale, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Philadelphia Hand to Shoulder Clinic, Philadelphia, Pennsylvania
  - Jefferson Rehabilitation, Philadelphia, Pennsylvania
  - Philadelphia Hand to Shoulder Center, Rockledge, Pennsylvania
  - Jefferson Rehabilitation, Torresdale, Pennsylvania
  - Jefferson Rehabilitation, Warminster, Pennsylvania
  - Jefferson Rehabilitation, Willow Grove, Pennsylvania
  - Philadelphia Hand to Shoulder Center, Willow Grove, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided
Pending discussion with TJU console.

DOCUMENTS (1):
  • Informed Consent Form (2023-08-16): https://cdn.clinicaltrials.gov/large-docs/65/NCT06025565/ICF_000.pdf